CLINICAL TRIAL: NCT05757661
Title: Effectiveness of Focal Vibration on the Performance of Amateur Athletes
Brief Title: Focal Vibration on the Performance of Amateur Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Jacobo Rodríguez Sanz, Principal investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIS-2022-05
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Vibration; Exposure; Sports Physical Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focal Vibration Group (Experimental)
  Interventions: Other: Focal Vibration
- Sham Group (Sham Comparator)
  Interventions: Other: Sham Group

INTERVENTIONS:
Other: Focal Vibration — A single 30-minute focal vibration procedure will be performed on both quadriceps with the V-Plus Wintecare® machine.
  Three channels will be used on the muscle bellies of the rectus anterior, vastus internus and vastus externus. The positioning of the vibration heads will be done with straps designed by the manufacturer to keep the vibration focus stable on the muscle belly.
  The configuration of the vibration program will be in an automatic mode of 10 seconds of vibration and 3 seconds of rest to avoid the coupling of the mechanoreceptors. The frequency used will be between 60 Hz to 150 Hz with a power of 80%.
  Arms: Focal Vibration Group
Other: Sham Group — The same procedure of the intervention group will be performed but without the focal vibration head contacting the skin (sham). A sufficient space will be left between the head and the headgear so that the vibration does not touch the skin.
  Arms: Sham Group

SUMMARY:
Focal vibration is an adjustable instrument, which has the ability to apply vibration to a specific point at different hertz, powers and rhythms. The use of general or focused vibration is not new in the rehabilitation or sports field. Vibration is intended to stimulate neuromuscular uses to produce involuntary and additional contractions of muscle tissue, indirectly causing an increase in strength or muscle mass , improved fall prevention, mobility and bone consolidation. This type of device has been used both in athletes and in patients with chronic diseases or in intensive care units. There are studies that use vibration in critically ill patients because it is a safe and feasible intervention for dependent patients. One of the advantages of focal vibration is that it can be used in both unloading and loading, which allows a wide range of adaptation to each patient, even simultaneously during a training activity.

The aim of the present study is to evaluate the effectiveness of a focal vibration treatment on strength, jumping and running speed in national federated athletes who perform sprinting and jumping in their sports practice.

A sample will be recruited during the months of April to September, estimating a sample of 70 total subjects (35 subjects in the vibration group and 35 subjects in the vibration placebo group).

Patients will receive a single treatment and assessments will be performed on the same day.

The focal vibration group will receive a 30-minute quadriceps intervention. 3 channels will be used on the muscle bellies of the rectus anterior, vastus internus and vastus externus. The vibration program configuration will be in an automatic mode of 10 seconds of vibration 3 seconds of rest to avoid mechanoreceptor coupling. The frequency used will be between 60 Hz to 150 Hz with a power of 80%. The placebo group will perform the same treatment as the intervention group but without the focal vibration head contacting the skin (placebo). A sufficient space will be left between the head and the headgear so that the vibration does not touch the skin as shown in previous studies.

A V-Plus machine (Wintecare S.A.) will be used for the vibration treatment. For the assessment measurements, a surface electromyograph, a force measurement dynamometer, the MyJump2 application for jump assessment and two photoelectric cells for sprint measurement will be used.

DETAILED DESCRIPTION:
Focal vibration is an adjustable instrument, which has the ability to apply vibration to a specific point at different hertz, powers and rhythms. The use of general or focused vibration is not new in the rehabilitation or sports field. Vibration is intended to stimulate neuromuscular uses to produce involuntary and additional contractions of muscle tissue, indirectly causing an increase in strength or muscle mass , improved fall prevention, mobility and bone consolidation. This type of device has been used both in athletes and in patients with chronic diseases or in intensive care units. There are studies that use vibration in critically ill patients because it is a safe and feasible intervention for dependent patients. One of the advantages of focal vibration is that it can be used in both unloading and loading, which allows a wide range of adaptation to each patient, even simultaneously during a training activity.

As mentioned above, focal vibration has had good results in increasing muscle mass; however, there is no study that has assessed whether focal vibration generates immediate improvements in the performance of functional tests such as jumping, maximum strength or running speed.

Different studies have observed improved activation of muscle fibers after applying global and/or focal vibration; however, it is not known whether activation is maintained in more functional gestures that require maximum effort (such as jumping or sprinting) in trained individuals.

The aim of the present study is to evaluate the effectiveness of a focal vibration treatment on strength, jumping and running speed in national federated athletes who perform sprinting and jumping in their sports practice.

A sample will be recruited during the months of April to September, estimating a sample of 70 total subjects (35 subjects in the vibration group and 35 subjects in the vibration placebo group).

Patients will receive a single treatment and assessments will be performed on the same day.

The focal vibration group will receive a 30-minute quadriceps intervention. 3 channels will be used on the muscle bellies of the rectus anterior, vastus internus and vastus externus. The vibration program configuration will be in an automatic mode of 10 seconds of vibration 3 seconds of rest to avoid mechanoreceptor coupling. The frequency used will be between 60 Hz to 150 Hz with a power of 80%. The placebo group will perform the same treatment as the intervention group but without the focal vibration head contacting the skin (placebo). A sufficient space will be left between the head and the headgear so that the vibration does not touch the skin as shown in previous studies.

A V-Plus machine (Wintecare S.A.) will be used for the vibration treatment. For the assessment measurements, a surface electromyograph, a force measurement dynamometer, the MyJump2 application for jump assessment and two photoelectric cells for sprint measurement will be used.

ELIGIBILITY:
Inclusion Criteria:

* Athletes between 18 and 30 years of age (athletics and field sports such as soccer, basketball, rugby... that may involve sprinting) federated and competing in university or national amateur leagues that perform sprinting and jumping in their sports practice.
* Active participation in regional, national or international competitions.
* Study participants must have signed the informed consent form in order to evaluate their inclusion in the study.

Exclusion Criteria:

* Volunteers who have suffered a sports injury during the last two months or are unable to perform physical activity.
* Not understanding the information provided by the therapist.
* Participate in other research studies.
* Being under a pharmacological medical treatment that may interfere with the measures, such as treatment with anticonvulsants, antidepressants, etc.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in 30 meters sprint (seconds) | Baseline(immediately before intervention) and post intervention (immediately after intervention)
  Photoelectric cells will be used to measure the time required to complete a 30-meter sprint.
Changes in electromyographic activity during sprint (μ/v) | Baseline(immediately before intervention) and post intervention (immediately after intervention)
  The mean electromyographic activity of the quadriceps musculature during sprint will be measured with The mDurance® system device (mDurance Solutions SL, Granada, Spain).

SECONDARY OUTCOMES:
Countermovement jump (cm) | Baseline(immediately before intervention) and post intervention (immediately after intervention)
  A bipodal jump will be performed and measured with the validated application "MyJump 2".
Changes in electromyographic activity during countermovement jump (μ/v) | Baseline(immediately before intervention) and post intervention (immediately after intervention)
  The mean electromyographic activity of the quadriceps musculature during the jump will be measured with The mDurance® system device (mDurance Solutions SL, Granada, Spain).
Changes in isometric leg extension (Newtons) | Baseline(immediately before intervention) and post intervention (immediately after intervention)
  A precision dynamometer (Microfeet II) will be used and the maximum force during an isometric contraction of this musculature during 5 seconds of the quadriceps will be analyzed.
Changes in electromyographic activity during isometric leg extension (μ/v) | Baseline(immediately before intervention) and post intervention (immediately after intervention)
  The mean electromyographic activity of the quadriceps musculature during the isometric leg extension will be measured with The mDurance® system device (mDurance Solutions SL, Granada, Spain).

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain